CLINICAL TRIAL: NCT04310800
Title: Ligation of Intersphincteric Fistula Tract Versus Ligation of the Intersphincteric Fistula Tract Plus a Bioprosthetic Anal Fistula Plug Procedure in Patients With Transsphincteric Anal Fistula: Multicenter Prospective Randomized Trial
Brief Title: LIFT-plug vs LIFT, a RCT Trial
Acronym: LIFT 02
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhen Jun Wang (Other)
Collaborators: The Second Artillery General Hospital (Other); Peking University Third Hospital (Other); Beijing Anorectal Hospital (Other); Beijing Luhe Hospital (Other); Beijing Shuyi Hospital (Other); People's Hospital of Beijing Daxing District (Other)
Responsible Party: Sponsor-Investigator, Zhen Jun Wang, Professor, Beijing Chao Yang Hospital
Organization: Beijing Chao Yang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LIFT-plug 2020; 2018-1-2032 (Other Grant/Funding Number: the Capital Health Research and Development of Special)
Record Dates: First submitted 2020-03-13; First posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Anal Fistula; LIFT-plug; Healing Rate; Anal Function
Keywords: anorectal fistula; LIFT-plug; complications of treatment; healing rate; anal function
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Who Masked: Participant
Masking Description: Randomization was performed on the day before surgery through sealed opaque envelopes containing the surgical method. The study was approved by the institutional review boards of the 7 hospitals.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LIFT-plug (Experimental): The LIFT-plug procedure was performed as followings. A portion of the fistula tract was excised from ei¬ther end within the intersphincteric space. One porcine small-intestine submucosa extracellular matrix plug was soaked in saline for 5-10 min, then placed into the intersphincteric groove and pulled through the curetted tract to the external opening. The plug was secured with a figure-of-eight 3/0 absorbable suture to the fistula opening in the external sphincter and ligated. Excess plug protruding from the external opening was trimmed flush with the skin without fixation. The wound was loosely closed with 2-3 interrupted 3/0 absorbable sutures.
  Interventions: Procedure: LIFT-plug technique
- LIFT (Experimental): The LIFT procedure was performe as followings. The curvilinear incision and dissection of the intersphincteric tract were made as in the LIFT-plug technique. After the tract was isolated, the tract was doubly-ligated and suture-ligated with absorbable sutures as close as possible to the lateral margin of the internal anal sphincter and the medial margin of the external anal sphincter. The tract was then divided between the two sutures. A portion of the fistula tract was excised after ligation of ei¬ther end within the intersphincteric space. The medial ligature was very close to the internal opening, and nearly obliterated the internal opening. The external opening was then enlarged to allow adequate drainage. The internal and external sphincters were then re-approximated, and the skin was closed loosely with interrupted 3/0 absorbable suture.
  Interventions: Procedure: LIFT-plug technique

INTERVENTIONS:
Procedure: LIFT-plug technique — Small-intestine submucosa extracellular matrix plug was soaked in saline for 5-10 min, then placed into the intersphincteric groove and pulled through the curetted tract to the external opening. The plug was secured with a figure-of-eight 3/0 absorbable suture to the fistula opening in the external sphincter and ligated. Excess plug protruding from the external opening was trimmed flush with the skin without fixation. The wound was loosely closed with 2-3 interrupted 3/0 absorbable sutures

SUMMARY:
To validate the effect of Ligation of Intersphincteric Fistula Tract (LIFT) Versus LIFT-plug procedure for Anal Fistula Repair in 7 medical centers

DETAILED DESCRIPTION:
The management of trans-sphincteric anal fistulae of cryptoglandular origin is challenging. The ideal management is to effectively heal the fistula without compromising continence, avoid fistula recurrence, and quick recovery. Ligation of the intersphincteric fistula tract (LIFT) and LIFT reinforced with a bioprosthetic graft (BioLIFT) are two recently reported procedures that showed improved healing results. In the LIFT, Rojanasakul et al proposed to identify the fistula tract in the intersphincteric space and subsequent division and ligation of the tract, and the primary healing rate was 94.4%. The following studies reported slightly lower results, but the recurrence rate was as high as 18% to 28%. Ellis et al subsequently described a modified LIFT procedure (BioLIFT procedure) in which a bioprosthetic was placed in the intersphincteric plane to reinforce the closure of the fistula tract (BioLIFT procedure), and yielded a healing rate of 94% in 31 patients who had a minimum of 1 year of follow-up after their last treatment. The investigators modified the LIFT procedure by combining LIFT with the technique of anal fistula plug. The bioprosthetic plug was placed into the fistula tract through the opening in the external sphincter to the external opening in the skin after LIFT procedure. The present study was designed to assess the preliminary results of LIFT-Plug technique prospectively. The purpose of this study is to validate the effect of Ligation of Intersphincteric Fistula Tract (LIFT) Versus LIFT-plug procedure for Anal Fistula Repair in 7 medical centers.

ELIGIBILITY:
Inclusion Criteria:

* High transsphincteric fistula (involving > 30% of the external anal sphincter)
* Age between 18 and 70 years
* Chronic anal fistula with fistula tracts no more than 2
* No active sepsis or abscess

Exclusion Criteria:

* Fistulas with active inflammation or purulence
* Fistulas related to tumor, Crohn's disease, tuberculosis or acquired immune deficiency syndrome
* Poorly controlled diabetes with fasting blood-glucose > 8mmol/L
* Preexisting incontinence
* Multiple fistula tracts > 2
* Fasting blood-glucose ≥ 8mmol/L
* Allergic or contraindication for the use of animal protein
* Pregnant women
* Expected life less than 6 months
* With anorectal abscess
* Serious liver (Child-Pugh C) and chronic kidney disease (CKD) stage 3

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Healing rate | 6 months postoperatively
  the healing rate of two groups in 6 months postoperatively
healing time | 6 months postoperatively
  the wound healing time from operation to healing

SECONDARY OUTCOMES:
anal function | 5 days, 2 weeks, 1 months, 3 months and 1 year postoperatively
  wexner score
pain score postoperatively | 5 days, 2 weeks, 1 months, 3 months and 1 year postoperatively
  visual analog scale scores

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Beijing Anorectal Hospital, Beijing, Beijing Municipality
  - Beijing Luhe Hospital, Beijing, Beijing Municipality
  - Beijing shunyi district hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Rocket force general hospital, Beijing, Beijing Municipality
  - Beijing Chaoyang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing daxing district people's hospital, Beijing

IPD SHARING:
Plan to Share IPD: Undecided